CLINICAL TRIAL: NCT03909763
Title: Combination of Danazole With Berberine in the Treatment of ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZXH81470343
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Corticosteroid-resistant or Relapsed ITP
Keywords: corticosteroid-resistant or relapsed ITP; Danazole; berberine
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Berberine; Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Berberine plus danazol (Experimental): Berberine plus danazol group
  Interventions: Drug: Berberine plus danazol

INTERVENTIONS:
Drug: Berberine plus danazol — Oral BBR (0.3g thrice daily) plus oral danazol (200 mg twice daily) for 16 weeks
  Other Names: HangZhou Mingsheng of China

SUMMARY:
A prospective, multicenter, open-label, Phase II, single arm, trial performed in 6 departments of hematology in China

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an autoimmune disorder characterized by low platelet count and mucocutaneous bleeding. Approximately one-third of ITP patients fail to respond to first-line therapies. In addition, a certain amount of the patients relapse and require further therapy after one or more treatment strategies (e.g., thrombopoietin receptor agonists or rituximab). The optimal second-line treatment remains a challenge.Berberine (BBR), an isoquinoline alkaloid derived from plants, is widely used as a nonprescription drug to treat diarrhea. Our previous data demonstrated that gut microbiota dysbiosis may contribute to the development of corticosteroid-resistant ITP. BBR may correct corticosteroid-resistance by modulating the gut microbiota structure, thus being a novel potential second-line candidate to treat ITP. Importantly, the potential clinical benefits of BBR have already been evaluated in various studies using human subjects, and it has been shown to be safe. Danazol is an attenuated androgen that has successfully been used in the treatment of ITP. Considering the side-effects of a regular dose of danazol and that BBR and danazol share disparate mechanisms in the treatment of ITP, we hypothesized that the combination of these two agents might be a promising option to maximize efficacy while minimizing adverse effects. Therefore, we aimed to evaluate the long-term efficacy and safety of berberine plus danazol in patients with corticosteroid-resistant or relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed immune thrombocytopenic purpura (ITP) newly diagnosed
2. Platelet count less than 30×109/L on two occasions or Platelets above 30×109/L combined with bleeding manifestation
3. Subject is ≥ 18 years and ≤80years
4. Subject has signed and dated written informed consent.
5. Fertile patients must use effective contraception during treatment and observational period
6. Negative pregnancy test

Exclusion Criteria:

1. Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL
2. Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an aspartate aminotransaminase or alanine aminotransferase level > 3×upper limit of normal
3. Have a New York Heart Classification III or IV heart disease
4. Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures
5. Have active hepatitis B or hepatitis C infection
6. Have a HIV infection
7. Have active infection requiring antibiotic therapy within 7 days prior to study entry
8. Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug
9. Previous treatment with rituximab
10. Previous splenectomy
11. Had previous or concomitant malignant disease
12. Not willing to participate in the study.
13. Expected survival of < 2 years
14. Intolerant to murine antibodies
15. Immunosuppressive treatment within the last month
16. Connective tissue disease
17. Autoimmune hemolytic anemia
18. Patients currently involved in another clinical trial with evaluation of drug treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University of people's hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Berberine Plus Danazol
Started | 55
Completed | 45
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Berberine Plus Danazol
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 45 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Count of Participants That Achieved 6-month Sustained Response
Description: 6-month sustained response defined as platelet count of 30×10⁹/L or more and at least a doubling of baseline platelet count (partial response (PR)), or a platelet count of 100×10⁹/L or more and the absence of bleeding without rescue medication(complete response (CR))
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Berberine Plus Danazol
Number analyzed (Participants) | 45
Participants | 28

2. Secondary Outcome: the Count of Participants That Had Adverse Events
Description: any adverse events/serious adverse events associated with study drugs and bleeding events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Berberine Plus Danazol
Number analyzed (Participants) | 45
Participants
  Adverse events associated with study drugs | 4
  Bleeding events | 1
  No adverse events | 40

3. Secondary Outcome: the Count of Participants That Achieved Initial Response
Description: Initial response by day 28. Initial response includes partial response (PLT of 30×10⁹/L or more and at least a doubling of baseline platelet count) and complete response (PLT of 100×10⁹/L or more and the absence of bleeding without rescue medication).
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Berberine Plus Danazol
Number analyzed (Participants) | 45
Participants | 21

4. Secondary Outcome: DOR
Description: duration of response (DOR)
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Berberine Plus Danazol
Number analyzed (Participants) | 45
months | 9.2 (10.731)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Berberine Plus Danazol
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Berberine Plus Danazol (N=45)
Intracranial bleeding (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berberine Plus Danazol (N=45)
seborrheic dermatitis (Endocrine disorders) | 3 (3)
androgenetic alopecia (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03909763/Prot_SAP_000.pdf